CLINICAL TRIAL: NCT05964075
Title: A Randomized Controlled Trial to Assess the Safety and Efficiency of a Self-Contained Sampling Device /disposable Bronchoscope System Versus Usual SampLing Procedure.
Brief Title: RASECAL-Bronchoscopic Ambusampler
Acronym: Rasecal
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RASECAL Study
Record Dates: First submitted 2023-04-18; First posted 2023-07-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Prospective, multi-centre, open labelled, 1:1randomized controlled study.

DETAILED DESCRIPTION:
1. Patients admitted to ICU with acute respiratory failure, requiring mechanical ventilation with, suspected or confirmed COVID-19.
2. Patients admitted to ICU with acute respiratory failure due to a condition other than COVID-19, requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

(All are required)

* Clinicians experienced in performing bronchoscopies (i.e. bronchoscopists should have performed a minimum 5 bronchoscopies in mechanically ventilated patients and a minimum of 5 bronchoscopies in a simulated or practice setting).
* Clinicians who have undergone the online product-training module for the use of the Ambu Bronchosampler, with self-certification documented.
* Clinicians who have simulated the online product training module using an Ambu Bronchosampler and Ambu Ascope4 a minimum of 5 times in a practice setting and have self-certified.

Population

* Patients ≥ 18 years old
* Patients on mechanical ventilation with Acute respiratory failure for >4h
* Patients eligible for a clinically indicated bronchoscopy with fluid sampling. Patient information has been explained and verbal or written consent has been obtained

Exclusion Criteria:

Investigators

* Investigators who have not completed product training in aScope BronchoSampler by online and hands-on from Ambu product specialists or an experienced user from the site.
* Investigators with experience in < 5 self-verified simulated fluid sampling procedures using the Ambu BronchoSampler 4.8.2 Population
* Clinician concern regarding safety of bronchoscopy
* Involved study personal not available to perform the procedure and enroll the patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring clinical bronchoscopy
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Comparison of two sampling pots | 1month
  Can the Ambu Bronchosampler improve safety versus usual standard care by reducing the risk of spillage or disconnection of the sampling system during a procedure?

CONTACTS AND LOCATIONS:
Overall Officials: Damon 0 Foster, 0, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital NHSFT, London, United Kingdom